CLINICAL TRIAL: NCT01833403
Title: Metabolomic Analysis of Hepatic Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1211M23881
Record Dates: First submitted 2013-04-10; First posted 2013-04-16 (Estimated); Results first posted 2015-06-16 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: bariatric surgery, l; liver insulin resistance,
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Glucose Clamp Technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Measurement of insulin sensitivity (Other): All participants will undergo a hyperinsulinemic-euglycemic clamp to measure insulin sensitivity
  Interventions: Other: Hyperinsulinemic-euglycemic clamp

INTERVENTIONS:
Other: Hyperinsulinemic-euglycemic clamp — Subject will received 6,6 2H2 Glucose prior and during a 4 hr hyperinsulinemic-euglycemic clamp to characterize hepatic insulin resistance prior to bariatric surgery
  --------------------------------------------------------------------------------
  Other Names: glucose clamp

SUMMARY:
This is a pilot study to show that it is possible to identify the specific types of fats in blood, adipose tissue, and liver tissue. The study doctors hope to use the analysis of these fats to learn more about nonalcoholic fatty liver disease (NFLD). Nonalcoholic fatty liver disease is the accumulation of fat in the liver of people who have minimal alcohol exposure. Nonalcoholic Fatty Liver Disease is associated with obesity and insulin resistance, and predicts development of Type 2 Diabetes. The study doctors are interested in looking at the relationship between liver fat and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible to participate in the study will be:

1. Adults over age 18;
2. Patients enrolled in the bariatric surgery clinic who are planning to undergo and have insurance approval for bariatric surgery;
3. Insulin sensitive (based on HOMA-IR calculated from screening labs) OR insulin resistant (based on HOMA-IR and or personal history of diet controlled diabetes)
4. Able and willing to give informed consent.

Exclusion Criteria

The following will exclude subjects from study participation:

1. Clinically significant medical issues outside of diabetes (eg, pregnancy, cardiovascular disease, uncontrolled pulmonary disease). If female and of child bearing potential, a pregnancy test will be performed and confirmed negative prior to participation in the study and prior to the scheduled glucose clamp procedure.
2. A history of hematologic (platelets <100 x107/L), hepatic (liver function tests [LFTs] >2X upper limit of normal), renal (Creatinine >1.5 mg/dL), pulmonary/ cardiac abnormalities (ie, abnormal electrocardiogram [EKG]).
3. Use of anti-diabetes medication, anticoagulants, or medication that might alter lipids. If the subject has a history of diabetes, it should be controlled by diet alone.
4. Inflammatory or celiac intestinal disease;
5. Untreated thyroid disease;
6. Excessive alcohol use, illicit drug use, or active untreated psychiatric disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Chow, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Data too small (n=4) to be shared publicly, although we will share deidentified data upon case-by-case request

RESULTS

PARTICIPANT FLOW:
Groups:
- Hyperinsulinemic-euglycemic Clamp: hyperinsulinemic-euglycemic clamp
  Hyperinsulinemic-euglycemic clamp: Subject will received 6,6 2H2 Glucose prior and during a 4 hr hyperinsulinemic-euglycemic clamp to characterize hepatic insulin resistance prior to bariatric surgery
  --------------------------------------------------------------------------------
  Glucose
Period: Overall Study
Arm/Group | Hyperinsulinemic-euglycemic Clamp
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hyperinsulinemic-euglycemic Clamp
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 4
insulin sensitivity [Mean (Standard Deviation); unit: HOMA IR] | 3.55 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: m value
Arm/Group | Hyperinsulinemic-euglycemic Clamp
Number analyzed (Participants) | 4
m value | 8 (2)
Statistical Analysis 1: Comparison: Hyperinsulinemic-euglycemic Clamp; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Primary Outcome: Insulin Sensitivity
Description: Insulin sensitivity was assessed during the euglycemic/hyperglycemic clamp test. Insulin-mediated glucose uptake (M-value) was calculated as the mean glucose requirement during the 150-180 minute interval of the clamp
Time Frame: 1 month
Measure: Mean (Standard Error); unit: mg glucose /kg FFM/min
Groups:
- Measurement of Insulin Sensitivity: All participants will undergo a hyperinsulinemic-euglycemic clamp to measure insulin sensitivity
  Hyperinsulinemic-euglycemic clamp: Subject will received 6,6 2H2 Glucose prior and during a 4 hr hyperinsulinemic-euglycemic clamp to characterize hepatic insulin resistance prior to bariatric surgery
  --------------------------------------------------------------------------------
Arm/Group | Measurement of Insulin Sensitivity
Number analyzed (Participants) | 4
mg glucose /kg FFM/min | 8.5 (2)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Hyperinsulinemic-euglycemic Clamp
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No